CLINICAL TRIAL: NCT01304797
Title: A Phase 1, Multi-Center, Open-Label, Dose-Escalation, Safety, and Pharmacokinetic Clinical Study of Intravenously Administered MM-302 Monotherapy and in Combination With Trastuzumab With or Without Cyclophosphamide in Patients With Advanced HER2 Positive Breast Cancer
Brief Title: Safety and Pharmacokinetic Study of MM-302 in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-302-02-01-01
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: MM302; Breast Cancer; Locally advanced/unresectable; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — gancotamab; Trastuzumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MM-302 (Experimental)
  Interventions: Drug: MM-302 Monotherapy
- MM-302 in Combination with Trastuzumab (Experimental)
  Interventions: Drug: MM-302 in combination with trastuzumab
- MM-302 in Combination with Trastuzumab q3w (Experimental)
  Interventions: Drug: MM-302 in combination with trastuzumab q3w
- MM-302 in Combination with Trastuzumab and Cyclophosphamide (Experimental)
  Interventions: Drug: MM-302 in combination with trastuzumab and cyclophosphamide

INTERVENTIONS:
Drug: MM-302 Monotherapy — Escalating doses of MM-302 as a single agent
  Arms: MM-302
Drug: MM-302 in combination with trastuzumab — Escalating MM-302 at an every 4 week dosing schedule, while the dose of trastuzumab is fixed at an every 2 week dosing schedule
  Other Names: Herceptin
  Arms: MM-302 in Combination with Trastuzumab
Drug: MM-302 in combination with trastuzumab q3w — Escalating MM-302 at an every 3 week dosing schedule, while the dose of trastuzumab is fixed at an every 3 week dosing schedule
  Other Names: herceptin
  Arms: MM-302 in Combination with Trastuzumab q3w
Drug: MM-302 in combination with trastuzumab and cyclophosphamide — Escalating MM-302 at an every 3 week dosing schedule, while the dose of trastuzumab and cyclophosphamide is fixed at an every 3 week dosing schedule
  Other Names: herceptin; cytoxan; neosar
  Arms: MM-302 in Combination with Trastuzumab and Cyclophosphamide

SUMMARY:
This study is a Phase 1 and pharmacologic open-label dose-escalation trial using a "3+3" design. Successive cohorts of three or more patients will be treated at escalating doses until a maximum tolerated dose is identified. Once the maximum tolerated dose is identified, an Expansion Cohort will be enrolled at that dose to further characterize safety and pharmacologic endpoints. Additional arms will be enrolled to explore the combination of MM-302 with trastuzumab or trastuzumab plus cyclophosphamide in patients with advanced HER2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced/unresectable or metastatic breast cancer
* Eighteen years of age or above
* Able to understand and sign an informed consent (or have a legal representative who is able to do so)
* Measurable disease according to RECIST v1.1
* ECOG Performance Score of 0 or 1
* Adequate bone marrow, hepatic, renal and cardiac function
* Willing to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of MM-302

Exclusion Criteria:

* Patients for whom potentially curative anticancer therapy is available
* Active infection or fever > 38.5°C during screening visits or on the first scheduled day of dosing
* Symptomatic CNS disease
* Known hypersensitivity to any of the components of MM-302 or who have had hypersensitivity reactions to fully human monoclonal antibodies
* Received other recent antitumor therapy
* Pregnant or breast feeding
* Patients with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The severity and the number of adverse events related to escalating doses of the MM-302. | 12 months
The severity and the number of adverse events related to escalating doses of the MM-302 in combination with trastuzumab with or without cyclophosphamide | 12 months

SECONDARY OUTCOMES:
Objective response rate of MM-302 | 12 months
The pharmacokinetics of MM-302 as determined by measuring AUC, Tmax and Cmax | 12 months
Immunogenicity of MM-302 by confirming whether MM-302 elicits an immune response or not | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - University of Indiana, Indianapolis, Indiana
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri

REFERENCES:
- [Derived] Lee H, Shields AF, Siegel BA, Miller KD, Krop I, Ma CX, LoRusso PM, Munster PN, Campbell K, Gaddy DF, Leonard SC, Geretti E, Blocker SJ, Kirpotin DB, Moyo V, Wickham TJ, Hendriks BS. 64Cu-MM-302 Positron Emission Tomography Quantifies Variability of Enhanced Permeability and Retention of Nanoparticles in Relation to Treatment Response in Patients with Metastatic Breast Cancer. Clin Cancer Res. 2017 Aug 1;23(15):4190-4202. doi: 10.1158/1078-0432.CCR-16-3193. Epub 2017 Mar 15. PMID 28298546